CLINICAL TRIAL: NCT06213506
Title: A Phase IIa Observer-blind, Randomized, Controlled, Age-de-escalation, Single Center Interventional Study to Evaluate the Safety, Reactogenicity, and Immune Response of the GVGH iNTS Vaccine Against S. Typhimurium and S. Enteritidis, in Adults, Children and Infants, Including Dose-finding in Infants, in Africa
Brief Title: A Study on the Safety, Reactogenicity, and Immune Response to the GVGH iNTS-GMMA Vaccine Against Invasive Nontyphoidal Salmonella in Adults, Children, and Infants
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: European & Developing Countries Clinical Trials Partnership (Unknown); Kwame Nkrumah University of Science and Technology (Other); Pedvac iNTS consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 217218
Record Dates: First submitted 2023-12-19; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Salmonella Infections
Keywords: GVGH iNTS-GMMA vaccine; Safety; Reactogenicity; Immunogenicity; sub-Saharan Africa; African adults, children and infants; Age de-escalation; Dose escalation; Invasive nontyphoidal Salmonella
MeSH Terms: conditions — Salmonella Infections | interventions — Rubella Vaccine; Yellow Fever Vaccine; Vaccines, Combined; Pneumococcal Vaccines; Poliovirus Vaccine, Inactivated; MenACWY; Meningococcal Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Intervention Model Description: Data will be collected in an observer-blind manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (22):
- Adults_Dose C Group (Experimental): Adults 18-50 years of age, part of the safety cohort, randomized to receive 2 doses of the iNTS-GMMA Dose C vaccine at Day 1 and Day 57.
  Interventions: Biological: iNTS-GMMA Dose C
- Adults_Control Group (Active Comparator): Adults 18-50 years of age, part of the safety cohort, randomized to receive 1 dose of the MenACWY vaccine at Day 1 and 1 dose of Placebo at Day 57.
  Interventions: Biological: MenACWY; Drug: Placebo
- Children_Dose B Group (Experimental): Children 24-59 months of age, part of the safety cohort, randomized to receive 2 doses of the iNTS-GMMA Dose B vaccine at Day 1 and Day 57.
  Interventions: Biological: iNTS-GMMA Dose B
- Children_Control B Group (Active Comparator): Children 24-59 months of age, part of the safety cohort, randomized to receive 2 doses of the MenACWY vaccine at Day 1 and Day 57.
  Interventions: Biological: MenACWY
- Children_Dose C Group (Experimental): Children 24-59 months of age, part of the safety cohort, randomized to receive 2 doses of the iNTS-GMMA Dose C vaccine at Day 1 and Day 57.
  Interventions: Biological: iNTS-GMMA Dose C
- Children_Control C Group (Active Comparator): Children 24-59 months of age, part of the safety cohort, randomized to receive 2 doses of the MenACWY vaccine at Day 1 and Day 57.
  Interventions: Biological: MenACWY
- Infants_9M_Dose A Group (Experimental): Infants 9 months of age, part of the safety cohort, randomized to receive 3 doses of the iNTS-GMMA Dose A vaccine at Day 1, Day 85 and Day 169. These infants also receive an Expanded Program on Immunization (EPI) vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the first study intervention administration occurring at Day 1, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: iNTS-GMMA Dose A
- Infants_9M_Control A Group (Active Comparator): Infants 9 months of age, part of the safety cohort, randomized to receive 2 doses of the MenACWY vaccine at Day 1 and Day 85 and 1 dose of the DTPaHBV-IPV+Hib vaccine at Day 169. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the first study intervention administration occurring at Day 1, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: MenACWY; Combination Product: DTPa-HBV-IPV+Hib
- Infants_9M_Dose B Group (Experimental): Infants 9 months of age, part of the safety cohort, randomized to receive 3 doses of the iNTS-GMMA Dose B vaccine at Day 1, Day 85 and Day 169. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the first study intervention administration occurring at Day 1, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: iNTS-GMMA Dose B
- Infants_9M_Control B Group (Active Comparator): Infants 9 months of age, part of the safety cohort, randomized to receive 2 doses of the MenACWY vaccine at Day 1 and Day 85 and 1 dose of the DTPaHBV-IPV+Hib vaccine at Day 169. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the first study intervention administration occurring at Day 1, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: MenACWY; Combination Product: DTPa-HBV-IPV+Hib
- Infants_9M_Dose C Group (Experimental): Infants 9 months of age, part of the safety cohort, randomized to receive 3 doses of the iNTS-GMMA Dose C vaccine at Day 1, Day 85 and Day 169. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the first study intervention administration occurring at Day 1, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: iNTS-GMMA Dose C
- Infants_9M_Control C Group (Active Comparator): Infants 9 months of age, part of the safety cohort, randomized to receive 2 doses of the MenACWY vaccine at Day 1 and Day 85 and 1 dose of the DTPaHBV-IPV+Hib vaccine at Day 169. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the first study intervention administration occurring at Day 1, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: MenACWY; Combination Product: DTPa-HBV-IPV+Hib
- Infants_6W_Dose A Group (Experimental): Infants 6 weeks of age, part of the safety cohort, randomized to receive 3 doses of the iNTS-GMMA Dose A vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the third study intervention administration occurring at Day 232, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: iNTS-GMMA Dose A
- Infants_6W_Control A Group (Active Comparator): Infants 6 weeks of age, part of the safety cohort, randomized to receive 3 doses of the MenACWY vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). To allow completion of the vaccination schedule a fourth dose of the MenACWY vaccine is administered after the trial ends, as per the licensed indication and in private vaccination settings. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the third study intervention administration occurring at Day 232, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: MenACWY
- Infants_6W_Dose B Group (Experimental): Infants 6 weeks of age, part of the safety cohort, randomized to receive 3 doses of the iNTS-GMMA Dose B vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the third study intervention administration occurring at Day 232, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: iNTS-GMMA Dose B
- Infants_6W_Control B Group (Active Comparator): Infants 6 weeks of age, part of the safety cohort, randomized to receive 3 doses of the MenACWY vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). To allow completion of the vaccination schedule a fourth dose of the MenACWY vaccine is administered after the trial ends, as per the licensed indication and in private vaccination settings. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the third study intervention administration occurring at Day 232, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: MenACWY
- Infants_6W_Dose C Group (Experimental): Infants 6 weeks of age, part of the safety cohort, randomized to receive 3 doses of the iNTS-GMMA Dose C vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the third study intervention administration occurring at Day 232, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: iNTS-GMMA Dose C
- Infants_6W_Control C Group (Active Comparator): Infants 6 weeks of age, part of the safety cohort, randomized to receive 3 doses of the MenACWY vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). To allow completion of the vaccination schedule a fourth dose of the MenACWY vaccine is administered after the trial ends, as per the licensed indication and in private vaccination settings. These infants also receive an EPI vaccination with Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine at 28 days after the third study intervention administration occurring at Day 232, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: MenACWY
- Infants_6W_Dose A_2 Group (Experimental): Infants 6 weeks of age, part of the dose-finding cohort, randomized to receive 3 doses of the iNTS-GMMA Dose A vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). These infants also receive an EPI vaccination with the following vaccines: Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine administered concomitantly during the last iNTS-GMMA administration at Day 232, and the pentavalent vaccine (DTPwHepB-Hib), the Pneumococcal conjugate vaccine, and the inactivated polio vaccine administered at the same time, at 6, 10 and 14 weeks of age, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: Pentavalent vaccine; Biological: Pneumococcal vaccine; Biological: Inactivated polio vaccine; Biological: iNTS-GMMA Dose A
- Infants_6W_Dose B_2 Group (Experimental): Infants 6 weeks of age, part of the dose-finding cohort, randomized to receive 3 doses of the iNTS-GMMA Dose B vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). These infants also receive an EPI vaccination with the following vaccines: Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine administered concomitantly during the last iNTS-GMMA administration at Day 232, and the pentavalent vaccine (DTPwHepB-Hib), the Pneumococcal conjugate vaccine, and the inactivated polio vaccine administered at the same time, at 6, 10 and 14 weeks of age, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: Pentavalent vaccine; Biological: Pneumococcal vaccine; Biological: Inactivated polio vaccine; Biological: iNTS-GMMA Dose B
- Infants_6W_Dose C_2 Group (Experimental): Infants 6 weeks of age, part of the dose-finding cohort, randomized to receive 3 doses of the iNTS-GMMA Dose C vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). These infants also receive an EPI vaccination with the following vaccines: Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine administered concomitantly during the last iNTS-GMMA administration at Day 232, and the pentavalent vaccine (DTPwHepB-Hib), the Pneumococcal conjugate vaccine, and the inactivated polio vaccine administered at the same time, at 6, 10 and 14 weeks of age, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: Pentavalent vaccine; Biological: Pneumococcal vaccine; Biological: Inactivated polio vaccine; Biological: iNTS-GMMA Dose C
- Infants_6W_Control_2 Group (Active Comparator): Infants 6 weeks of age, part of the dose-finding cohort, randomized to receive 3 doses of the MenACWY vaccine at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase). To allow completion of the vaccination schedule a fourth dose of the MenACWY vaccine is administered after the trial ends, as per the licensed indication and in private vaccination settings. These infants also receive an EPI vaccination with the following vaccines: Measles and Rubella Vaccine (MR-VAC) and Yellow Fever (YF) vaccine administered concomitantly during the last study intervention administration at Day 232, and the pentavalent vaccine (DTPw-HepB-Hib), the Pneumococcal conjugate vaccine, and the inactivated polio vaccine administered at the same time, at 6, 10 and 14 weeks of age, at the local EPI vaccination centers, and not part of the current clinical trial.
  Interventions: Biological: Measles and Rubella vaccine; Biological: Yellow Fever vaccine; Biological: Pentavalent vaccine; Biological: Pneumococcal vaccine; Biological: Inactivated polio vaccine; Biological: MenACWY

INTERVENTIONS:
Biological: Measles and Rubella vaccine — Measles and Rubella vaccine is administered to study participants, as part of an Expanded Program on Immunization (EPI) vaccination at the local EPI vaccination centers, and not part of the current clinical trial, as follows: - at 28 days after the first study intervention administration (occurring at Day 1) to infants in the Infants_9M_Dose A, Infants_9M_Control A, Infants_9M_Dose B, Infants_9M_Control B, Infants_9M_Dose C and Infants_9M_Control C groups. - at 28 days after the third study intervention administration (occurring at Day 232) to infants in Infants_6W_Dose A, Infants_6W_Control A, Infants_6W_Dose B, Infants_6W_Control B, Infants_6W_Dose C and Infants_6W_Control C groups. - at Day 232, concomitantly during the last study intervention administration to infants in Infants_6W_Dose A_2, Infants_6W_Dose B_2, Infants_6W_Dose C_2 and Infants_6W_Control_2 groups.
  Other Names: MR-VAC
  Arms: Infants_6W_Control A Group; Infants_6W_Control B Group; Infants_6W_Control C Group; Infants_6W_Control_2 Group; Infants_6W_Dose A Group; Infants_6W_Dose A_2 Group; Infants_6W_Dose B Group; Infants_6W_Dose B_2 Group; Infants_6W_Dose C Group; Infants_6W_Dose C_2 Group; Infants_9M_Control A Group; Infants_9M_Control B Group; Infants_9M_Control C Group; Infants_9M_Dose A Group; Infants_9M_Dose B Group; Infants_9M_Dose C Group
Biological: Yellow Fever vaccine — Yellow Fever vaccine is administered to study participants, as part of an Expanded Program on Immunization (EPI) vaccination at the local EPI vaccination centers, and not part of the current clinical trial, as follows: - at 28 days after the first study intervention administration (occurring at Day 1) to infants in the Infants_9M_Dose A, Infants_9M_Control A, Infants_9M_Dose B, Infants_9M_Control B, Infants_9M_Dose C and Infants_9M_Control C groups. - at 28 days after the third study intervention administration (occurring at Day 232) to infants in Infants_6W_Dose A, Infants_6W_Control A, Infants_6W_Dose B, Infants_6W_Control B, Infants_6W_Dose C and Infants_6W_Control C groups. - at Day 232, concomitantly during the last study intervention administration to infants in Infants_6W_Dose A_2, Infants_6W_Dose B_2, Infants_6W_Dose C_2 and Infants_6W_Control_2 groups.
  Arms: Infants_6W_Control A Group; Infants_6W_Control B Group; Infants_6W_Control C Group; Infants_6W_Control_2 Group; Infants_6W_Dose A Group; Infants_6W_Dose A_2 Group; Infants_6W_Dose B Group; Infants_6W_Dose B_2 Group; Infants_6W_Dose C Group; Infants_6W_Dose C_2 Group; Infants_9M_Control A Group; Infants_9M_Control B Group; Infants_9M_Control C Group; Infants_9M_Dose A Group; Infants_9M_Dose B Group; Infants_9M_Dose C Group
Biological: Pentavalent vaccine — Pentavalent vaccine is administered, as part of an Expanded Program on Immunization (EPI) vaccination, at the local EPI vaccination centers, and not part of the current clinical trial, at 6, 10 and 14 weeks of age to infants in Infants_6W_Dose A_2, Infants_6W_Dose B_2, Infants_6W_Dose C_2 and Infants_6W_Control_2 groups.
  Other Names: DTPw-HepB-Hib
  Arms: Infants_6W_Control_2 Group; Infants_6W_Dose A_2 Group; Infants_6W_Dose B_2 Group; Infants_6W_Dose C_2 Group
Biological: Pneumococcal vaccine — Pneumococcal vaccine is administered, as part of an Expanded Program on Immunization (EPI) vaccination, at the local EPI vaccination centers, and not part of the current clinical trial, at 6, 10 and 14 weeks of age to infants in Infants_6W_Dose A_2, Infants_6W_Dose B_2, Infants_6W_Dose C_2 and Infants_6W_Control_2 groups.
  Arms: Infants_6W_Control_2 Group; Infants_6W_Dose A_2 Group; Infants_6W_Dose B_2 Group; Infants_6W_Dose C_2 Group
Biological: Inactivated polio vaccine — Inactivated polio vaccine is administered, as part of an Expanded Program on Immunization (EPI) vaccination, at the local EPI vaccination centers, and not part of the current clinical trial, at 6, 10 and 14 weeks of age to infants in Infants_6W_Dose A_2, Infants_6W_Dose B_2, Infants_6W_Dose C_2 and Infants_6W_Control_2 groups.
  Arms: Infants_6W_Control_2 Group; Infants_6W_Dose A_2 Group; Infants_6W_Dose B_2 Group; Infants_6W_Dose C_2 Group
Biological: iNTS-GMMA Dose C — -2 doses of iNTS-GMMA Dose C vaccine administered intramuscularly, at Day 1 and Day 57 to adults and children in the Adults_Dose C and Children_Dose C groups; -3 doses of iNTS-GMMA Dose C vaccine administered intramuscularly, at Day 1, Day 85 and Day 169 to infants in the Infants_9M_Dose C group, and at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase) to infants in the Infants_6W_Dose C and Infants_6W_Dose C_2 groups.
  Arms: Adults_Dose C Group; Children_Dose C Group; Infants_6W_Dose C Group; Infants_6W_Dose C_2 Group; Infants_9M_Dose C Group
Biological: iNTS-GMMA Dose B — -2 doses of iNTS-GMMA Dose B vaccine administered intramuscularly, at Day 1 and Day 57 to children in the Children_Dose B group; -3 doses of iNTS-GMMA Dose B vaccine administered intramuscularly, at Day 1, Day 85 and Day 169 to infants in the Infants_9M_Dose B group, and at Day 1, Day 57 (during the Priming phase) and Day at 232 (during the Booster phase) to infants in the Infants_6W_Dose B and Infants_6W_Dose B_2 groups.
  Arms: Children_Dose B Group; Infants_6W_Dose B Group; Infants_6W_Dose B_2 Group; Infants_9M_Dose B Group
Biological: iNTS-GMMA Dose A — 3 doses of iNTS-GMMA Dose A vaccine administered intramuscularly, at Day 1, Day 85 and Day 169 to infants in the Infants_9M_Dose A group, and at Day 1, Day 57 (during the Priming phase) and Day at 232 (during the Booster phase) to infants in the Infants_6W_Dose A and Infants_6W_Dose A_2 groups.
  Arms: Infants_6W_Dose A Group; Infants_6W_Dose A_2 Group; Infants_9M_Dose A Group
Biological: MenACWY — -1 dose of MenACWY vaccine administered intramuscularly at Day 1 to adults in the Adults_Control group; -2 doses of MenACWY vaccine administered intramuscularly at Day 1 and Day 57 to children in the Children_Control B and Children_Control C groups, and at Day 1 and Day 85 to infants in the Infants_9M_Control A, Infants_9M_Control B and Infants_9M_Control C groups; -3 doses of MenACWY vaccine administered intramuscularly at Day 1, Day 57 (during the Priming phase) and at Day 232 (during the Booster phase) to infants in the Infants_6W_Control A, Infants_6W_Control B, Infants_6W_Control C and Infants_6W_Control_2 groups. A 4th dose of MenACWY vaccine is administered after the trial ends, to infants in the aforementioned study groups, as per the licensed indication and in private vaccination settings.
  Other Names: Menveo
  Arms: Adults_Control Group; Children_Control B Group; Children_Control C Group; Infants_6W_Control A Group; Infants_6W_Control B Group; Infants_6W_Control C Group; Infants_6W_Control_2 Group; Infants_9M_Control A Group; Infants_9M_Control B Group; Infants_9M_Control C Group
Combination Product: DTPa-HBV-IPV+Hib — 1 dose of DTPa-HBV-IPV+Hib vaccine administered intramuscularly at Day 169 to infants in the Infants_9M_Control A, Infants_9M_Control B and Infants_9M_Control C groups.
  Other Names: Infanrix hexa
  Arms: Infants_9M_Control A Group; Infants_9M_Control B Group; Infants_9M_Control C Group
Drug: Placebo — 1 dose of Placebo administered intramuscularly at Day 57 to adults in the Adults_Control group.
  Arms: Adults_Control Group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, and immune response of the GlaxoSmithKline (GSK) Vaccines Institute for Global Health (GVGH) invasive nontyphoidal Salmonella-generalized modules for membrane antigens (iNTS-GMMA) candidate vaccine against S. Typhimurium and S. Enteritidis with an age de-escalation and dose escalation approach in African population, starting with adults (18-50 years of age), then on children (24-59 months of age) and finally to infants (9 months and 6 weeks of age). Infants are the target for primary vaccination from 6 weeks of age.

DETAILED DESCRIPTION:
The study will be conducted in two stages:

Stage 1: Age De-escalation from Adults to Children and Infants

* Adult participants will receive either iNTS-GMMA Dose C (high) or a control vaccine intramuscularly on Day 1 and Day 57.
* Child participants will receive either Dose B (medium) or Dose C (high) of the candidate vaccine or the control on Day 1 and Day 57.
* Infant participants (9 months of age) will receive either Dose A (low), Dose B (medium), or Dose C (high) of the candidate vaccine or the control on Day 1, Day 85, and Day 169.
* Infant participants (6 weeks of age) will receive either Dose A (low), Dose B (medium), or Dose C (high) of the candidate vaccine or the control on Day 1, Day 85 (Priming phase), and Day 232 (Booster phase).

Stage 2: Dose-finding in Infants of 6 weeks of age

-Infants (6 weeks of age) will receive one of the three dose levels (Dose A [low], Dose B [medium], or Dose C [high]) of the candidate vaccine or the control on Day 1, Day 85 (Priming phase), and Day 232 (Booster phase).

ELIGIBILITY:
Inclusion criteria:

All participants (adults, children, infants at 9 months of age and infants at 6 weeks of age) will be enrolled in the clinical site in Ghana and must satisfy ALL the following criteria at study entry:

* Participants and/or participants' parent(s)/Legally Acceptable Representative(s) (LAR), who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the participant/parent(s)/LAR(s) of the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history, clinical examination, and laboratory investigations.
* Participants satisfying screening requirements.
* Participants negative for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C.

Adult participants must satisfy ALL the following criteria at study entry:

* A male or female between and including 18 and 50 years of age at the time of the first study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant:

has practiced adequate contraception for 1 month prior to study intervention administration, and:

* has a negative pregnancy test on the day of study intervention administration, and
* has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.

The Ghana card will be used as source document to verify the ages for the adults.

Child participants must satisfy ALL the following criteria at study entry:

* A male or female between and including 24 and 59 months of age at the time of the first study intervention administration.
* Previously completed routine childhood vaccinations to the best knowledge of the participant's parent(s)/LAR's.
* Born after a gestation period of ≥37 weeks.

Infant participants must satisfy ALL the following criteria at study entry:

* A male or female 6 weeks or 9 months of age at the time of the first study intervention administration.
* Born after a gestation period of ≥37 weeks.
* Born to a mother seronegative for HIV, hepatitis B virus and hepatitis C virus.

The Road to Health Chart will be used as source document to confirm the ages for the children and infants.

Exclusion criteria:

Medical conditions

* Known exposure to S. Typhimurium or S. Enteritidis during the period starting at birth for infants and children, and at 3 years for adults, as documented by patient records
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Hypersensitivity, including allergy, to medicinal products or medical equipment whose use is foreseen in this study.
* Progressive, unstable, or uncontrolled clinical conditions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Major congenital defects, as assessed by the investigator.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease and/or fever at the time of enrollment (fever is defined as temperature ≥ 38.0°C).
* Recurrent history or uncontrolled neurological disorders or seizures.
* Any clinically significant hematological and/or biochemical laboratory abnormality.
* Undernutrition defined as WHO Z-score less than -2 SD.
* Malaria infection defined as the presence of asexual parasites in the blood.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* History of receiving any investigational iNTS or GMMA vaccines in the participant's life.
* Use of any investigational or non-registered product other than the study interventions during the period beginning 30 days before the first dose of study interventions, or their planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 14 days before each dose and ending 28 days after the last dose of study interventions administration, with the exception of flu vaccines and vaccines administered as part of a public health vaccination campaign.
* A vaccine not foreseen by the study protocol administered during the period starting at 14 days before the first dose and ending 14 days after the last dose of study interventions administration for live vaccines or 7 days in case of inactivated vaccines*, with the exception of flu vaccines or COVID-19 vaccine which may be considered on a case-by-case basis.

  * If emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is organized by public health authorities outside the routine immunization program, the time period described above can be reduced if, provided it is used according to the local governmental recommendations and Sponsor is notified.

Under such circumstances, a participant may be considered eligible for study enrollment and/or study intervention administration after the appropriate window for delay has passed and inclusion/exclusion criteria have been re-checked, and if the participant is confirmed to be eligible.

* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives from birth (for infant 6 weeks of age) or during the period starting 3 months before the administration of the first dose of study intervention(s) or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose(s) up to the end of the study. For corticosteroids, this will mean prednisone equivalent greater than or equal to (>=) 20 mg/day for adult participants/ >= 0.5 mg/kg/day with maximum of 20 mg/day for pediatric participants (infants and children). Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (vaccine, drug and device).

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of/current chronic alcohol consumption and/or drug abuse. This will be decided at the discretion of the investigator.
* Any study personnel or their immediate dependents, family, or household members.
* Child in care.

Ages: 6 Weeks to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 516 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) in infants 6 weeks of age part of the dose-finding cohort | At Day 85 (28 days after the second study intervention administration)
  Anti-Salmonella Typhimurium (S. Typhimurium) O antigen (Ag) total IgG and anti-Salmonella Enteritidis (S. Enteritidis) OAg total IgG GMCs are assessed.
Percentage of adult participants 18-50 years of age with solicited administration site events | During 7 days after the first study intervention administration occurring at Day 1
  The solicited administration site events are pain, redness and swelling.
Percentage of adult participants 18-50 years of age with solicited administration site events | During 7 days after the second study intervention administration occurring at Day 57
  The solicited administration site events are pain, redness and swelling.
Percentage of adult participants 18-50 years of age with solicited systemic events | During 7 days after the first study intervention administration occurring at Day 1
  The solicited systemic events are fever, headache, myalgia, arthralgia and fatigue. Fever is defined as axillary temperature higher than or equal to (>=) 38.0 degrees Celsius (°C)/100.4 degrees Fahrenheit (°F).
Percentage of adult participants 18-50 years of age with solicited systemic events | During 7 days after the second study intervention administration occurring at Day 57
  The solicited systemic events are fever, headache, myalgia, arthralgia and fatigue. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of adult participants 18-50 years of age with unsolicited adverse events (AEs) | During 28 days after the first study intervention administration occurring at Day 1
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of adult participants 18-50 years of age with unsolicited adverse events (AEs) | During 28 days after the second study intervention administration occurring at Day 57
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of adult participants 18-50 years of age with serious adverse events (SAEs) | From first study intervention administration (Day 1) up to the end of study participation (Day 85)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, or results in abnormal pregnancy outcomes.
Percentage of adult participants 18-50 years of age with adverse events (AEs) leading to withdrawal from the study or discontinuation of study intervention | From first study intervention administration (Day 1) up to the end of study participation (Day 85)
  An AE is any untoward medical occurrence (an unfavorable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. Any AEs that lead to discontinuation of study intervention and/or the study are considered under this outcome measure.
Percentage of adult participants 18-50 years of age with deviations from reference ranges l or baseline values for hematological, renal and hepatic panel test results | At Day 8 (7 days after the first study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of adult participants 18-50 years of age with deviations from reference ranges or baseline values for hematological, renal and hepatic panel test results | At Day 64 (7 days after the second study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of child participants 24-59 months of age with solicited administration site events | During 7 days after the first study intervention administration occurring at Day 1
  The solicited administration site events are pain, redness and swelling.
Percentage of child participants 24-59 months of age with solicited administration site events | During 7 days after the second study intervention administration occurring at Day 57
  The solicited administration site events are pain, redness and swelling.
Percentage of child participants 24-59 months of age with solicited systemic events | During 7 days after the first study intervention administration occurring at Day 1
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of child participants 24-59 months of age with solicited systemic events | During 7 days after the second study intervention administration occurring at Day 57
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of child participants 24-59 months of age with unsolicited AEs | During 28 days after the first study intervention administration occurring at Day 1
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of child participants 24-59 months of age with unsolicited AEs | During 28 days after the second study intervention administration occurring at Day 57
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of child participants 24-59 months of age with serious adverse events (SAEs) | From first study intervention administration (Day 1) up to the end of study participation (Day 85)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity or any other situation based on appropriate medical or scientific judgement.
Percentage of child participants 24-59 months of age with AEs leading to withdrawal from the study or discontinuation of study intervention | From first study intervention administration (Day 1) up to the end of study participation (Day 85)
  An AE is any untoward medical occurrence (an unfavorable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. Any AEs that lead to discontinuation of study intervention and/or the study are considered under this outcome measure.
Percentage of child participants 24-59 months of age with deviations from reference ranges or baseline values for hematological, renal and hepatic panel test results | At Day 8 (7 days after the first study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of child participants 24-59 months of age with deviations from reference ranges or baseline values for hematological, renal and hepatic panel test results | At Day 64 (7 days after the second study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of infant participants 9 months of age with solicited administration site events | During 7 days after the first study intervention administration occurring at Day 1
  The solicited administration site events are pain, redness and swelling.
Percentage of infant participants 9 months of age with solicited administration site events | During 7 days after the second study intervention administration occurring at Day 85
  The solicited administration site events are pain, redness and swelling.
Percentage of infant participants 9 months of age with solicited administration site events | During 7 days after the third study intervention administration occurring at Day 169
  The solicited administration site events are pain, redness and swelling.
Percentage of infant participants 9 months of age with solicited systemic events | During 7 days after the first study intervention administration occurring at Day 1
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness, and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of infant participants 9 months of age with solicited systemic events | During 7 days after the second study intervention administration occurring at Day 85
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness, and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of infant participants 9 months of age with solicited systemic events | During 7 days after the third study intervention administration occurring at Day 169
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness, and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of infant participants 9 months of age with unsolicited adverse events (AEs) | During 28 days after the first study intervention administration occurring at Day 1
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of infant participants 9 months of age with unsolicited adverse events (AEs) | During 28 days after the second study intervention administration occurring at Day 85
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of infant participants 9 months of age with unsolicited adverse events (AEs) | During 28 days after the third study intervention administration occurring at Day 169
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of infant participants 9 months of age with serious adverse events (SAEs) | From first study intervention administration (Day 1) up to the end of study participation (Day 337)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity or any other situation based on appropriate medical or scientific judgement.
Percentage of infant participants 9 months of age with adverse events (AEs) leading to withdrawal from the study or discontinuation of study intervention | From first study intervention administration (Day 1) up to the end of study participation (Day 337)
  An AE is any untoward medical occurrence (an unfavorable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. Any AEs that lead to discontinuation of study intervention and/or the study are considered under this outcome measure.
Percentage of infant participants 9 months of age with deviations from reference range or baseline values for hematological, renal and hepatic panel test results | At Day 8 (7 days after the first study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of infant participants 9 months of age with deviations from reference range or baseline values for hematological, renal and hepatic panel test results | At Day 92 (7 days after the second study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of infant participants 9 months of age with deviations from reference range or baseline values for hematological, renal and hepatic panel test results | At Day 176 (7 days after the third study intervention administration)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of infant participants 6 weeks of age with solicited administration site events | During 7 days after the first study intervention administration occurring at Day 1 in the Priming phase
  The solicited administration site events are pain, redness and swelling.
Percentage of infant participants 6 weeks of age with solicited administration site events | During 7 days after the second study intervention administration occurring at Day 57 in the Priming phase
  The solicited administration site events are pain, redness and swelling.
Percentage of infant participants 6 weeks of age with solicited systemic events | During 7 days after the first study intervention administration occurring at Day 1 in the Priming phase
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness, and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of infant participants 6 weeks of age with solicited systemic events | During 7 days after the second study intervention administration occurring at Day 57 in the Priming phase
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness, and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F.
Percentage of infant participants 6 weeks of age with unsolicited adverse events (AEs) | During 28 days after the first study intervention administration occurring at Day 1 in the Priming phase
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of infant participants 6 weeks of age with unsolicited adverse events (AEs) | During 28 days after the second study intervention administration occurring at Day 57 in the Priming phase
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of infant participants 6 weeks of age with SAEs | From first study intervention administration (Day 1) up to 28 days after second study intervention (Day 85)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity or any other situation based on appropriate medical or scientific judgement.
Percentage of infant participants 6 weeks of age with adverse events (AEs) leading to MR-VAC administration withdrawal from the study or discontinuation of study intervention | From first study intervention administration (Day 1) up to 28 days after second study intervention (Day 85)
  An AE is any untoward medical occurrence (an unfavorable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. Any AEs that lead to discontinuation of study intervention and/or the study are considered under this outcome measure.
Percentage of infant participants 6 weeks of age with deviations from reference ranges or baseline values for hematological, renal, and hepatic panel test results | At Day 8 (7 days after the first study intervention administration) in the Priming phase
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of infant participants 6 weeks of age with deviations from reference ranges or baseline values for hematological, renal, and hepatic panel test results at Day 64 | At Day 64 (7 days after the second study intervention administration) in the Priming phase
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.

SECONDARY OUTCOMES:
Percentage of infant participants 6 weeks of age with solicited administration site events | During 7 days after the third study intervention administration occurring at Day 232 in the Booster phase
  The solicited administration site events are pain, redness and swelling.
Percentage of infant participants 6 weeks of age with solicited systemic events | During 7 days after the third study intervention administration occurring at Day 232 in the Booster phase
  The solicited systemic events are fever, irritability/fussiness, loss of appetite, drowsiness, and vomiting. Fever is defined as axillary temperature >= 38.0 °C/100.4 degrees °F
Number of infant participants 6 weeks of age with unsolicited AEs | During 28 days after the third study intervention administration occurring at Day 232 in the Booster phase
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of infant participants 6 weeks of age with SAEs | From 28 days after the second study intervention administration (Day 85) up to end of study participation (Day 400)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity or any other situation based on appropriate medical or scientific judgement.
Percentage of infant participants 6 weeks of age with adverse events (AEs) leading to withdrawal from the study or discontinuation of study intervention | From 28 days after the second study intervention administration (Day 85) up to end of study participation (Day 400)
  An AE is any untoward medical occurrence (an unfavorable /unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. Any AEs that lead to discontinuation of study intervention and/or the study are considered under this outcome measure.
Percentage of infant participants 6 weeks of age with deviations from reference ranges or baseline values for hematological, renal, and hepatic panel test results | At Day 239 (7 days after the study intervention administration) in the Booster phase
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) in infants 6 weeks of age dose finding cohort | At Day 260 (28 days after the booster study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG GMCs are assessed.
Anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) in adult participants 18-50 years of age | At Days 1 and 57 (before each study intervention administration) and at Days 29 and 85 (28 days after each study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG GMCs are assessed.
Anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) in child participants 24-59 months of age | At Days 1 and 57 (before each study intervention administration) and at Days 29 and 85 (28 days after each study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG GMCs are assessed.
Anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) in infant participants 9 months of age | At Days 1, 85 and 169 (before each study intervention administration) and at Days 29, 113 and 197 (28 days after each study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG GMCs are assessed.
Anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) geometric mean concentrations (GMCs) in infant participants 6 weeks of age | At Days 1, 57 and 232 (before each study intervention administration) at Days 29, 85 and 260 (28 days after each study intervention administration) and at Day 239 (7 days after the third study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG GMCs are assessed.
Percentage of adult participants 18-50 years of age achieving, for each antigen (Ag), at least a 2-fold and 4-fold rise in anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) antibody concentration | At Days 29 and 85 (28 days after each study intervention administration) compared to Day 1 (baseline, prior to first study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgGantibody concentrations are assessed.
Percentage of child participants 24-59 months of age achieving, for each antigen (Ag), at least a 2-fold and 4-fold rise in anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) antibody concentration | At Days 29 and 85 (28 days after each study intervention administration) compared to Day 1 (baseline, prior to first study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG antibody concentrations are assessed.
Percentage of infant participants 9 months of age achieving, for each antigen (Ag), at least a 2-fold and 4-fold rise in anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) antibody concentration | At Days 29, 113 and 197 (28 days after each study intervention administration) compared to Day 1 (baseline, prior to first study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG antibody concentrations are assessed.
Percentage of infant participants 6 weeks of age achieving, for each antigen (Ag), at least a 2-fold and 4-fold rise in anti-invasive nontyphoidal Salmonella (iNTS) serotype specific immunoglobulin G (IgG) antibody concentration | At Days 29, 85 and 260 (28 days after each study intervention administration) and at Day 239 (7 days after the third study intervention administration) compared to Day 1 (baseline, prior to first study intervention administration)
  Anti-S. Typhimurium OAg total IgG and anti-S. Enteritidis OAg total IgG antibody concentrations are assessed.
Anti-Hepatitis B surface (HBs) antigen (Ag) geometric mean concentrations (GMCs), in a subset of infant participants 6 weeks of age (dose-finding cohort) | At Day 1 (before the first study intervention administration) and at Day 85 (28 days after the third pentavalent vaccine administration)
Anti-Hib polyribosylribitol phosphate (PRP) geometric mean concentrations (GMCs), in a subset of infant participants 6 weeks of age (dose-finding cohort) | At Day 1 (before the first study intervention administration) and at Day 85 (28 days after the third pentavalent vaccine administration)
Anti-measles immunoglobulin G (IgG) antibody geometric mean concentrations (GMCs), in a subset of infant participants 6 weeks of age (dose-finding cohort) | At Day 232 (before MR-VAC administration) and at Day 260 (28 days after MR-VAC administration)
Anti-rubella immunoglobulin G (IgG) antibody geometric mean concentrations (GMCs), in a subset of infant participants 6 weeks of age (dose-finding cohort) | At Day 232 (before MR-VAC administration) and at Day 260 (28 days after MR-VAC administration)
Percentage of a subset of infant participants 6 weeks of age (dose-finding cohort) achieving an anti-measles IgG antibody concentration of equal to or above (≥) 150 milli international units per milliliter (mIU/mL) and ≥ 200 mIU/mL | At Day 232 (before MR-VAC administration) and at Day 260 (28 days after MR-VAC administration)
Percentage of a subset of infant participants 6 weeks of age (dose finding cohort) achieving an anti-rubella IgG antibody concentration of ≥ 4 international units per milliliter (IU/mL) and ≥ 10 IU/mL | At Day 232 (before MR-VAC administration) and at Day 260 (28 days after MR-VAC administration)
Percentage of a subset of infant participants 6 weeks of age (dose finding cohort) achieving an anti-Hepatitis B IgG antibody concentration of ≥ 10 mIU/mL | At Day 1 (before the first study intervention administration) and at Day 85 (28 days after third pentavalent vaccine administration)
Percentage of a subset of infant participants 6 weeks of age (dose-finding cohort) achieving an anti-Hib polyribosylribitol phosphate (PRP) IgG antibody concentration of ≥ 0.15 microgram per milliliter (µg/mL) | At Day 1 (before the first study intervention administration) and at Day 85 (28 days after third pentavalent vaccine administration)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.